CLINICAL TRIAL: NCT01385748
Title: A Phase II, Multi-center, Randomised, Double-blind, Placebo-controlled Study Comparing the Efficacy and Safety of Clonidine Lauriad® 50 μg and 100 μg Mucoadhesive Buccal Tablet (MBT) Applied Once Daily to Those of Placebo in the Prevention and Treatment of Chemoradiation Therapy Induced Oral Mucositis in Patients With Head and Neck Cancer
Brief Title: Efficacy and Safety Study of Clonidine Lauriad® to Treat Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BA2009/28/01
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clonidine Lauriad® 50µg (Active Comparator): 50µg muco-adhesive buccal tablets, once de day, every day up to 8 weeks
  Interventions: Drug: Clonidine Lauriad® 50µg
- Clonidine Lauriad® 100µg (Active Comparator): 100µg muco-adhesive buccal tablets, once a day, every day up to 8 weeks
  Interventions: Drug: Clonidine Lauriad® 100µg
- Placebo Lauriad® (Placebo Comparator): Placebo muco-adhesive buccal tablets, once a day, every day up to 8 weeks
  Interventions: Drug: Placebo Lauriad®

INTERVENTIONS:
Drug: Clonidine Lauriad® 50µg — 50µg muco-adhesive buccal tablet once day every day up to 8 weeks
  Arms: Clonidine Lauriad® 50µg
Drug: Clonidine Lauriad® 100µg — 100µg muco-adhesive buccal tablets, once a day, every day up to 8 weeks
  Arms: Clonidine Lauriad® 100µg
Drug: Placebo Lauriad® — placebo muco-adhesive buccal tablets, once a day, every day up to 8 weeks
  Arms: Placebo Lauriad®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Clonidine Lauriad® to treat chemoradiation therapy induced severe oral mucositis in patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged > 18 years
* Suffering from a newly diagnosed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx histologically-confirmed and having undergone resective surgery
* Prior neoadjuvant chemotherapy allowed provided that, the patient did not experience a World Health Organization (WHO) grade > 2 oral mucositis during the neoadjuvant therapy.
* Patient eligible to receive concurrent chemo-radiation defined as:

  1. A continuous course of conventional external beam irradiation (IMRT eligible) with a minimum cumulative radiation dose of 50 Gy or a maximum of 70 Gy, based on a daily dosing between 1.8 and 2.2 Gy combined with platinum based chemotherapy on a weekly or tri-weekly cycles.
  2. Planned radiation treatment fields must include at least two oral tissue sites (among right or left buccal mucosa, floor of mouth, tongue, right or left soft palate) with each site receiving a total of 50 Gy or a maximum of 70 Gy. The radiation treatment plan will be reviewed by a designated radiation oncologist.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Screening laboratory tests:

  1. Haemoglobin ≥ 10g/dL
  2. Absolute neutrophil counts ≥ 1500 cells/mm3
  3. Platelets ≥ 100.000/mm3
  4. Conjugated bilirubin ≤ 2 times Upper Limit of Normal (ULN)
  5. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 ULN
  6. Negative serum pregnancy test
* Women of child bearing potential must have effective contraception method (oral or device)
* Signed written informed consent

Exclusion Criteria:

* Tumours of the lips, sinuses, salivary glands
* Prior radiation of the head and neck area
* Curative surgery less than 2 weeks or more than 15 weeks prior to the initiation of radiation therapy-chemotherapy (RT-CT)
* Presence of active infectious disease
* Presence of active oral infectious disease, including oropharyngeal candidiasis and/or orofacial herpes
* Presence of oral mucositis
* Known or suspected chronic viral diseases including HIV
* Systolic blood pressure < 100 mmHg and/or Diastolic blood pressure < 50 mmHg
* Recent stroke within the last 6 months
* Bradyarrhythmia (<60 b/min), including sinus node dysfunction or atrioventricular (AV) nodal conduction block 2nd or 3rd degree
* Subjects with orthostatic hypotension, defined by a decrease of systolic BP and/or diastolic BP above 20 mmHg when the patient stands up
* Renal insufficiency (creatinine blood level > 1.5ULN)
* Ongoing heavy alcohol consumption (>100g alcohol/day)
* Administration of any concomitant treatment likely to interfere with clonidine
* Known hypersensitivity to clonidine, history of allergy or intolerance to milk proteins or any other component of the product
* Presence of severe or uncontrolled depression
* Pregnant or breast-feeding women
* Inability to give informed consent or comply with study requirements
* Unable or unwilling to comply with follow-up visits
* Participation to a clinical trial within 30 days prior to randomization and during the entire duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bérangère Vasseur, MD, Study Director — Valerio Therapeutics
Locations (51):
- United States (19):
  - 21st Century Oncology of Arizona, Sun City, Arizona
  - Compassionate Cancer Care Medical Group, Corona, California
  - City of Hope, Duarte, California
  - California Cancer Associates for Researche and Excellence, Fresno, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - Central Coast Medical Oncology Corp., Santa Maria, California
  - Centura Health Research Center, Denver, Colorado
  - University of Connectcut Health Center, Farmington, Connecticut
  - AMPM Research Clinic, Miami, Florida
  - Barbara Ann Karmonos Cancer Hospital, Detroit, Michigan
  - Washington University School of medecine, St Louis, Missouri
  - Billings Clinic Montana, Billings, Montana
  - Winthrop University Hospital, Mineola, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center- Carolinas Health Care System, Charlotte, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Hershey Cancer Institut, Hershey, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (13):
  - Hospital Jean Minjoz, Besançon
  - CHU Morvan, Brest
  - Centre François Baclesse, Caen
  - Clinique Pasteur, Évreux
  - Centre Oscar Lambret, Lille
  - Clinique Chénieux, Limoges
  - Clinique Hartmann, Neuilly-sur-Seine
  - CH Lyon Sud, Pierre-Bénite
  - CHU La Milétrie, Poitiers
  - CHP St gregoire, Saint-Grégoire
  - Centre de Cancérologie Etienne-Dolet, Saint-Nazaire
  - Hôpital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Universitatsklinikum Erlangen Strahlenklinik, Erlangen
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Freiburg Klinik fur Strahlentherapie, Freiburg im Breisgau
  - Universitatsklinikum Leipzig, Leipzig
  - Paracelsius- Klinik, Osnabrück
- Hungary (4):
  - Bács-Kiskun Megyei Kórház Szegedi Tudományegyetem Általános Orvostudományi Kar Oktató Kórháza, Kecskemét, Nyíri U. 38
  - Jósa András Oktatókórház Egészségügyi Szolgáltató Nonprofit Kft., Nyíregyháza, Szent István Út 68
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc, Szentpéteri Kapu 72-76
  - Szent Imre Kórház, Budapest, Tétényi Út 12-16.
- Spain (9):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de La princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de octubre, Madrid
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Ramon y cajal, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital de Navarra, Pamplona
- Centre Hospitalier Universitaire, Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 183 participants were randomized from 6 countries during 4 years
Groups:
- Clonidine Lauriad® 50 µg: Clonidine Lauriad® 50 µg: 50 µg muco-adhesive buccal tablet once a day every day up to 8 weeks
- Clonidine Lauriad® 100 µg: Clonidine Lauriad® 100 µg: 100 µg muco-adhesive buccal tablets once a day every day up to 8 weeks
- Placebo Lauriad®: Placebo Lauriad®: placebo muco-adhesive buccal tablets once a day every day up to 8 weeks
Period: Overall Study
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad®
Started | 56 | 65 | 62
Completed | 41 | 51 | 49
Not Completed | 15 | 14 | 13
Not completed — Withdrawal by Subject | 7 | 4 | 5
Not completed — Noncompliance | 3 | 1 | 6
Not completed — Other | 1 | 7 | 1
Not completed — Adverse Event | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Clonidine Lauriad® 50 µg: Clonidine Lauriad® 50 µg: 50µg muco-adhesive buccal tablet once a day every day up to 8 weeks
- Clonidine Lauriad® 100 µg: Clonidine Lauriad® 100 µg: 100µg muco-adhesive buccal tablets once a day every day up to 8 weeks
- Placebo Lauriad®: Placebo Lauriad®: placebo muco-adhesive buccal tablets, once a day every day up to 8 weeks
- Total: Total of all reporting groups
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Total
Number analyzed (Participants) | 56 | 65 | 62 | 183
Age, Continuous [Median (Full Range); unit: years] | 58.8 [30 to 79] | 55.7 [22 to 75] | 56.6 [33 to 72] | 57.3 [22 to 79]
Age, Customized [Number; unit: participants]
  18 to 64 years | 43 | 58 | 50 | 151
  65 to 84 years | 13 | 7 | 12 | 32
  85 years and over | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 13 | 45
  Male | 40 | 49 | 49 | 138
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 53 | 61 | 59 | 173
  Other | 2 | 4 | 3 | 9
  Black | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 3 | 0 | 4
  United States | 0 | 2 | 4 | 6
  France | 31 | 27 | 30 | 88
  Switzerland | 0 | 2 | 0 | 2
  Germany | 10 | 11 | 10 | 31
  Spain | 14 | 20 | 18 | 52
Eastern Cooperative Oncology Group (ECOG) Score [Number; unit: participants] — ECOG performance status measured on 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self care, unable to carry out any work activities; 3=Capable of only limited self care, confined to bed/chair >50% of waking hours; 4=Completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=Dead.
  participants
    Score 0 | 42 | 41 | 42 | 125
    Score 1 | 14 | 22 | 20 | 56
    Score 2 | 0 | 2 | 0 | 2
Disease location [Number; unit: participants] — The location of the squamous cell carcinoma.
  participants
    Oral cavity | 26 | 37 | 30 | 93
    Oropharynx | 19 | 17 | 21 | 57
    Hypopharynx | 4 | 2 | 2 | 8
    Larynx | 4 | 6 | 5 | 15
    Oral cavity/oropharynx | 0 | 1 | 1 | 2
    Oral cavity/hypopharynx | 0 | 1 | 1 | 2
    Oral cavity/larynx | 1 | 0 | 0 | 1
    Oropharynx/hypopharynx | 2 | 1 | 1 | 4
    Oropharynx/larynx | 0 | 0 | 1 | 1
Disease location in oral cavity or oropharynx [Number; unit: participants] — Location of the squamous cell carcinoma (in oral cavity or oropharynx).
  participants
    Yes | 48 | 57 | 55 | 160
    No | 8 | 8 | 7 | 23
Mucosal irritation [Number; unit: participants] — The number of participants with mucosal irritation at baseline.
  participants
    Yes | 2 | 2 | 1 | 5
    No | 53 | 63 | 61 | 177
    Missing | 1 | 0 | 0 | 1
Tooth extraction [Number; unit: participants] — The number of participants having undergone tooth extraction at baseline.
  participants
    Yes | 30 | 32 | 32 | 94
    No | 25 | 32 | 30 | 87
    Missing | 1 | 1 | 0 | 2
Oral infection [Number; unit: participants] — The number of participants presenting with oral infection at baseline.
  participants
    Yes | 0 | 1 | 0 | 1
    No | 55 | 64 | 62 | 181
    Missing | 1 | 0 | 0 | 1
Prior surgery [Number; unit: participants] — The number of participants having undergone prior surgery.
  participants
    Yes | 55 | 64 | 61 | 180
    No | 1 | 1 | 1 | 3
Prior radiotherapy and/or chemotherapy [Number; unit: participants] — The number of participants previously treated with radiotherapy and/or chemotherapy.
  participants
    Yes | 54 | 62 | 61 | 177
    No | 2 | 3 | 1 | 6
Height [Median (Full Range); unit: cm] | 171 [153 to 182] | 170 [147 to 186] | 172 [145 to 190] | 171 [145 to 190]
Weight [Median (Full Range); unit: kg] | 71.3 [44 to 130] | 66 [43 to 123] | 69 [48 to 115] | 69 [43 to 130]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 23.7 [16.1 to 44.4] | 23.66 [16.8 to 40.3] | 23.33 [16.9 to 43.8] | 23.59 [16.1 to 44.4]
Disease duration [Median (Full Range); unit: months] — Duration of the squamous cell carcinoma at baseline.
  months | 2 [1 to 14] | 2 [1 to 99] | 2 [0 to 7] | 2 [0 to 99]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Radiation Dose at Which Severe Oral Mucositis (World Health Organization [WHO] Score ≥ 3) Was First Observed
Description: The primary endpoint planned in the protocol was the percentage of participants with an oral mucositis score greater than or equal to 3 using the WHO oral mucositis severity scale at a cumulative radiation dose of 50 Gy. This was modified by protocol amendment to the cumulative radiation dose at which a WHO score greater than or equal to 3 was first observed. This change was made to account for the fact that in real practice most patients receive a cumulative dose between 60 and 70 Gy. The presence of grade 3 or 4 oral mucositis was assessed twice weekly during the active phase (radiotherapy) by a trained radiation oncologist or an ear nose and throat specialist who took into account the field of radiation treatment. WHO score 3 = oral ulcers, liquid diet only; WHO score 4 = oral alimentation impossible. Each assessment was associated with the actual cumulative dose of radiotherapy.
Time Frame: 8 weeks
Population: The analysis was conducted on the Intent to treat population, defined as all participants who received at least one dose of investigational drug.
Measure: Median (95% Confidence Interval); unit: Cumulative radiation dose (Gy)
Groups:
- Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled: Pooled group of participants who received Clonidine Lauriad® 50 ug muco-adhesive buccal tablets or Clonidine Lauriad® 100 ug muco-adhesive buccal tablets once a day every day up to 8 weeks.
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 56 | 65 | 62 | 121
Cumulative radiation dose (Gy) | 66 [44 to NA] — NA indicates that the upper limit of the confidence interval was not reached. | 56 [44 to NA] — NA indicates that the upper limit of the confidence interval was not reached. | 48 [42 to 61.6] | 60 [48 to NA] — NA indicates that the upper limit of the confidence interval was not reached.
Statistical Analysis 1: Comparison: Clonidine Lauriad® 50 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.165, Log Rank; The log rank test at 5% significance level was used; Hazard Ratio (HR) = 0.677, 95% CI 2-sided [0.387 to 1.186]
Statistical Analysis 2: Comparison: Clonidine Lauriad® 100 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.421, Log Rank; The log rank test at 5% significance level was used; Hazard Ratio (HR) = 0.817, 95% CI 2-sided [0.495 to 1.35]
Statistical Analysis 3: Comparison: Placebo Lauriad® vs Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled; Test type: Superiority or Other; p = 0.211, Log Rank; The log rank test at 5% significance level was used; Hazard Ratio (HR) = 0.754, 95% CI 2-sided [0.484 to 1.175]

2. Secondary Outcome: At Least One Opioid Use (Class 3 Analgesic)
Description: Opioid use was recorded twice weekly during the active phase (radiotherapy)
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad®
Number analyzed (Participants) | 56 | 65 | 62
participants
  Missing | 2 | 1 | 0
  Yes | 23 | 30 | 30
  No | 31 | 34 | 32

3. Secondary Outcome: Opioid Use: Minimal Total Cumulative Dose Administered (Mean, Standard Deviation)
Description: Opioid use was recorded twice weekly for up to 8 weeks during the active phase (radiotherapy). The sum of non-missing total cumulative doses across all class 3 analgesics recorded for the considered participant is reported.
Time Frame: 8 weeks
Population: Participants with at least one use of an opioid during the active phase with evaluable data.
Measure: Mean (Standard Deviation); unit: morphine dose equivalent
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 20 | 24 | 29 | 44
morphine dose equivalent | 469.31 (633.51) | 415.49 (490.55) | 624.94 (958.81) | 439.95 (553.88)

4. Secondary Outcome: Opioid Use: Minimal Total Cumulative Dose Administered (Median, Range)
Description: as for outcome 3
Time Frame: 8 weeks
Population: Participants with at least one use of an opioid during the active phase with evaluable data.
Measure: Median (Full Range); unit: morphine dose equivalent
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 20 | 24 | 29 | 44
morphine dose equivalent | 183.6 [12 to 2249.1] | 174 [15 to 1804] | 215 [20 to 3672] | 178.65 [12 to 2249.1]
Statistical Analysis 1: Comparison: Clonidine Lauriad® 50 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.807, Wilcoxon (Mann-Whitney) — Significance threshold = 5%
Statistical Analysis 2: Comparison: Clonidine Lauriad® 100 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.971, Wilcoxon (Mann-Whitney) — Significance threshold = 5%

5. Secondary Outcome: Overall Survival
Description: After the end-of study visit, the investigator center collects OS follow-up data for each patient who has consented to participate in the follow-up data collection. the OS follow-up period was still ongoing at time of the primary analysis and ended in Nov 2016. The analysis was condicted on the ITT population. The overall survival was evaluate every 6 months after last subject completed in patients who has consented to participate .
Time Frame: 2 years
Population: The population for the 2-year OS follow-up was the ITT defined as all patients who received at least 1 dose of investigational drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 56 | 65 | 62 | 121
months | 47 [17.3 to NA] — NA indicate that the upper limit of the confidence interval was not reached | 58.8 [35.9 to NA] — NA indicate that the upper limit of the confidence interval was not reached | 41.8 [27.7 to NA] — NA indicate that the upper limit of the confidence interval was not reached | 58.8 [32.3 to NA] — NA indicate that the upper limit of the confidence interval was not reached

6. Other Pre Specified Outcome: Time to Onset of Severe Oral Mucositis
Description: Time to onset is the duration until first Severe Oral Mucositis. Severe Oral Mucositis was defined as a Grade 3 or Grade 4 score on the World Health Organization (WHO) oral mucositis severity scale. Participants were assessed twice weekly during the active phase (radiotherapy) by a trained radiation oncologist or an ear nose and throat specialist who took into account the field of radiation treatment. WHO score 3 = ulcers, extensive erythema, and the inability of the participant to swallow a solid diet; WHO score 4 = mucositis to the extent that alimentation was not possible.
Time Frame: 8 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 56 | 65 | 62 | 121
weeks | 6.4 [4.6 to NA] — NA indicates that the upper limit of the confidence interval was not reached. | 6 [4.6 to 8] | 5.1 [4.4 to 6.9] | 6.4 [5.1 to NA] — NA indicates that the upper limit of the confidence interval was not reached.
Statistical Analysis 1: Comparison: Clonidine Lauriad® 50 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.199, Log Rank — Significance threshold = 5%; Hazard Ratio (HR) = 0.698, 95% CI 2-sided [0.398 to 1.223]
Statistical Analysis 2: Comparison: Clonidine Lauriad® 100 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.424, Log Rank; Significance threshold = 5%; Hazard Ratio (HR) = 0.817, 95% CI 2-sided [0.493 to 1.353]
Statistical Analysis 3: Comparison: Placebo Lauriad® vs Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled; Test type: Superiority or Other; p = 0.235, Log Rank; Significance threshold = 5%; Hazard Ratio (HR) = 0.764, 95% CI 2-sided [0.489 to 1.193]

7. Other Pre Specified Outcome: The Maximum Severity of Oral Mucositis
Description: Participants were assessed using the World Health Organization (WHO) oral mucositis severity scale twice weekly during the active phase (radiotherapy) by a trained radiation oncologist or an ear nose and throat specialist who took into account the field of radiation treatment. The WHO scores were as follows: 0 = None; 1 = oral soreness, erythema; 2 = oral erythema, ulcers, solid diet tolerated; 3 = oral ulcers, liquid diet only; 4 = oral alimentation impossible. The maximum severity was the maximum score reported during the active phase.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 56 | 65 | 62 | 121
participants
  Grade 0 | 7 | 6 | 4 | 13
  Grade 1 | 9 | 7 | 9 | 16
  Grade 2 | 15 | 20 | 11 | 35
  Grade 3 | 17 | 20 | 30 | 37
  Grade 4 | 6 | 10 | 6 | 16
  No value during the concerned period | 2 | 2 | 2 | 4
Statistical Analysis 1: Comparison: Clonidine Lauriad® 50 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.176, Kruskal-Wallis; Significance threshold = 5%
Statistical Analysis 2: Comparison: Clonidine Lauriad® 100 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.61, Kruskal-Wallis; Significance threshold = 5%
Statistical Analysis 3: Comparison: Placebo Lauriad® vs Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled; Test type: Superiority or Other; p = 0.295, Kruskal-Wallis; Significance threshold = 5%

8. Other Pre Specified Outcome: The Overall Incidence of Grade 3/4 Mucositis During the Active Phase.
Description: The presence of grade 3 or 4 oral mucositis on the World Health Organization (WHO) oral mucositis severity scale was assessed twice weekly during the active phase (radiotherapy) by a trained radiation oncologist or an ear nose and throat specialist who took into account the field of radiation treatment. WHO score 3 = ulcers, extensive erythema, and the inability of the participant to swallow a solid diet; WHO score 4 = mucositis to the extent that alimentation was not possible.The number of participants with at least one Grade 3 or Grade 4 mucositis score during the active phase is reported.
Time Frame: 8 weeks
Population: Missing = participants without a WHO score during the active phase
Measure: Number; unit: participants
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 56 | 65 | 62 | 121
participants
  Missing | 2 | 2 | 2 | 4
  No | 31 | 33 | 24 | 64
  Yes | 23 | 30 | 36 | 53
Statistical Analysis 1: Comparison: Clonidine Lauriad® 50 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.063, Chi-squared — Significance threshold = 5%
Statistical Analysis 2: Comparison: Clonidine Lauriad® 100 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.169, Chi-squared
Statistical Analysis 3: Comparison: Placebo Lauriad® vs Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled; Test type: Superiority or Other; p = 0.064, Chi-squared; Significance threshold = 5%

9. Other Pre Specified Outcome: Salivary Flow Assessment Using the National Cancer Institute-Common Terminology Criteria (NCI-CTC) for Xerostomia: Time to First Grade 2 or Higher
Description: Salivary flow was assessed and scored by the investigator weekly using the NCI-CTC scale for xerostomia for up to 8 weeks during the active phase (radiotherapy). Time to appearance of Grade 2 or higher on the following 4-point scoring scale is reported: 0 = normal; 1 = symptomatic (dry or thick saliva) without significant dietary alteration (unstimulated saliva flow greater than 0.2 mL/minute); 2 = symptomatic and significant oral intake alterations (e.g. copious water, other lubricants, diet limited to purees and/or soft, moist foods) (unstimulated saliva 0.1 to 0.2 mL/minute); and 3 = symptoms leading to inability to adequately aliment orally, intravenous fluids, tube feedings, or total parenteral nutrition indicated (unstimulated saliva < 0.1 mL/minute).
Time Frame: 8 weeks
Population: Two of the 183 participants received study treatment but withdrew early without any safety assessments (1 in the clonidine Lauriad 50 μg group and 1 in the clonidine Lauriad 100 μg group). The safety population therefore included 181 participants.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Clonidine Lauriad® 100µg: Clonidine Lauriad® 100 µg: 100 µg muco-adhesive buccal tablets once a day every day up to 8 weeks
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 55 | 64 | 62 | 119
weeks | 6 [4.9 to 9.4] | 7.4 [6 to NA] — NA indicates that the upper limit of the confidence interval was not reached. | 5.1 [4.1 to 7.1] | 7.1 [5.7 to 9.4]
Statistical Analysis 1: Comparison: Clonidine Lauriad® 50 µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.388, Log Rank; Significance threshold = 5%; Hazard Ratio (HR) = 0.824, 95% CI 2-sided [0.484 to 1.401]
Statistical Analysis 2: Comparison: Clonidine Lauriad® 100µg vs Placebo Lauriad®; Test type: Superiority or Other; p = 0.054, Log Rank; Significance threshold = 5%; Hazard Ratio (HR) = 0.601, 95% CI 2-sided [0.357 to 1.012]
Statistical Analysis 3: Comparison: Placebo Lauriad® vs Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled; Test type: Superiority or Other; p = 0.102, Log Rank; Significance threshold = 5%; Hazard Ratio (HR) = 0.692, 95% CI 2-sided [0.444 to 1.078]

10. Other Pre Specified Outcome: Overall Treatment Compliance According to the Patient Diary
Description: All participants complete a daily questionnaire during the active phase (radiotherapy). Compliance = [ number of tablets / (end date of treatment - start date treatment + 1 ) ] * 100. The "number of tablets" is the number of days with a tablet applied and treatment start and end dates are the first and last dates of the patient diary with a tablet applied.
Time Frame: 8 weeks
Population: Participants with evaluable data.
Measure: Mean (Standard Deviation); unit: percentage of compliance
Arm/Group | Clonidine Lauriad® 50 µg | Clonidine Lauriad® 100 µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Number analyzed (Participants) | 55 | 64 | 62 | 119
percentage of compliance | 94.28 (8.23) | 93.12 (11.89) | 96.12 (5.59) | 93.66 (10.34)

ADVERSE EVENTS:
Description: Two of the 183 participants received study treatment but withdrew early without any safety assessments (1 in the clonidine Lauriad 50 μg group and 1 in the clonidine Lauriad 100 μg group). The safety population therefore included 181 participants.
Groups:
- Clonidine Lauriad® 50µg: Clonidine Lauriad® 50µg: 50µg muco-adhesive buccal tablet once a day every day up to 8 weeks
- Clonidine Lauriad® 100µg: Clonidine Lauriad® 100µg: 100µg muco-adhesive buccal tablets once a day every day up to 8 weeks
Arm/Group | Clonidine Lauriad® 50µg | Clonidine Lauriad® 100µg | Placebo Lauriad® | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled
Serious Adverse Events (participants affected / at risk) | 16/55 | 21/64 | 14/62 | 37/119
Other Adverse Events (participants affected / at risk) | 48/55 | 60/64 | 61/62 | 108/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine Lauriad® 50µg (N=55) | Clonidine Lauriad® 100µg (N=64) | Placebo Lauriad® (N=62) | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled (N=119)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemolytic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thromoboctyopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 4 (4) | 1 (1) | 0 (0) | 5 (5)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 3 (4) | 3 (4)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (5) | 3 (4) | 4 (6)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine Lauriad® 50µg (N=55) | Clonidine Lauriad® 100µg (N=64) | Placebo Lauriad® (N=62) | Clonidine Lauriad® Muco-adhesive Buccal Tablets Pooled (N=119)
Anaemia (Blood and lymphatic system disorders) | 9 (11) | 12 (16) | 11 (12) | 21 (27)
Leukopenia (Blood and lymphatic system disorders) | 10 (17) | 12 (19) | 8 (11) | 22 (36)
Neutropenia (Blood and lymphatic system disorders) | 7 (9) | 12 (15) | 8 (9) | 19 (24)
Lymphopenia (Blood and lymphatic system disorders) | 7 (10) | 8 (12) | 5 (10) | 15 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (13) | 6 (11) | 4 (4) | 12 (24)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 4 (5) | 3 (3) | 6 (7)
Nausea (Gastrointestinal disorders) | 29 (63) | 29 (41) | 44 (82) | 58 (104)
Dysphagia (Gastrointestinal disorders) | 18 (25) | 19 (23) | 29 (40) | 37 (48)
Dry mouth (Gastrointestinal disorders) | 22 (26) | 17 (21) | 17 (22) | 39 (47)
Vomiting (Gastrointestinal disorders) | 14 (26) | 15 (20) | 24 (32) | 29 (46)
Constipation (Gastrointestinal disorders) | 18 (20) | 17 (19) | 16 (16) | 35 (39)
Oral pain (Gastrointestinal disorders) | 16 (40) | 19 (70) | 16 (40) | 35 (110)
Dysgeusia (Gastrointestinal disorders) | 14 (15) | 11 (13) | 12 (12) | 25 (28)
Diarrhoea (Gastrointestinal disorders) | 7 (15) | 14 (22) | 13 (22) | 21 (37)
Odynophagia (Gastrointestinal disorders) | 7 (11) | 14 (21) | 8 (22) | 21 (32)
Stomatitis (Gastrointestinal disorders) | 6 (15) | 8 (18) | 8 (17) | 14 (33)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 6 (6) | 6 (6) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (3) | 5 (5) | 4 (5)
Aptyalism (Gastrointestinal disorders) | 1 (1) | 4 (5) | 3 (4) | 5 (6)
Salivary hypersecretion (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Asthenia (General disorders) | 9 (12) | 11 (14) | 14 (18) | 20 (26)
Mucosal inflammation (General disorders) | 8 (21) | 11 (19) | 6 (12) | 19 (40)
Pyrexia (General disorders) | 5 (5) | 10 (13) | 3 (3) | 15 (18)
Fatigue (General disorders) | 5 (5) | 5 (6) | 8 (10) | 10 (11)
General physical health deterioration (General disorders) | 3 (4) | 1 (2) | 2 (2) | 4 (6)
Pain (General disorders) | 3 (3) | 2 (3) | 4 (4) | 5 (6)
Oedema (General disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Oral candidiasis (Infections and infestations) | 3 (4) | 10 (11) | 9 (13) | 13 (15)
Fungal infection (Infections and infestations) | 2 (2) | 2 (2) | 7 (7) | 4 (4)
Candida infection (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 4 (4)
Radiation skin injury (Injury, poisoning and procedural complications) | 14 (24) | 22 (45) | 24 (35) | 36 (69)
Blood creatinine increased (Investigations) | 7 (7) | 3 (3) | 7 (7) | 10 (10)
Abnormal loss of weight (Metabolism and nutrition disorders) | 4 (4) | 11 (13) | 17 (19) | 15 (17)
Decreased appetite (Metabolism and nutrition disorders) | 6 (8) | 8 (11) | 5 (6) | 14 (19)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (3) | 4 (4)
Headache (Nervous system disorders) | 5 (6) | 2 (2) | 9 (9) | 7 (8)
Dizziness (Nervous system disorders) | 2 (2) | 6 (10) | 2 (3) | 8 (12)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1) | 3 (4) | 6 (6)
Renal failure (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 8 (8) | 8 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (6) | 3 (4) | 7 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3) | 6 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 11 (27) | 9 (17) | 8 (17) | 20 (44)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4) | 3 (3) | 8 (9)
Hypotension (Vascular disorders) | 3 (4) | 4 (4) | 1 (1) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less